CLINICAL TRIAL: NCT05662098
Title: Alternative Dosing And Prevention of Transfusions (ADAPT): A Prospective Study to Reduce Transfusion Requirements for Children With Sickle Cell Anemia Using Pharmacokinetics-based Hydroxyurea Dosing
Brief Title: Alternative Dosing And Prevention of Transfusions (ADAPT)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Jinja Regional Referral Hospital (JRRH), Sickle Cell Clinic, Jinja, Uganda (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADAPT
Record Dates: First submitted 2022-10-04; First posted 2022-12-22 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Sickle Cell Disease
Keywords: Pharmacokinetics; Hydroxyurea; Transfusion
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: ADAPT is a prospective cohort study at Jinja Regional Referral Hospital (JRRH) primarily to assess the effect of hydroxyurea on blood transfusion utilization and secondarily to determine the feasibility of PK-guided hydroxyurea dosing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): All participants will receive an individualized PK hydroxyurea assessment. Participants for whom the PK-process successfully generates a dose in the predicted treatment range of 15-35 mg/kg/day, will start on that personalized dose. Participants for whom the process does not generate a starting hydroxyurea dose in the predicted treatment range, due to potential pitfalls in lab draws, serum storage, sample processing, or hydroxyurea analysis, will start at a default dose of 20.0 ± 2.5 mg/kg/day. For all participants, the hydroxyurea dose will be adjusted as needed based on blood counts to establish the optimal dose. Where necessary, a weekly dosing average will be determined, so that treatment can occur solely with locally available and affordable 500mg hydroxyurea capsules.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — All participants will receive an individualized PK hydroxyurea assessment. Participants for whom the PK-process successfully generates a dose in the predicted treatment range of 15-35 mg/kg/day, will start on that personalized dose. Participants for whom the process does not generate a starting hydroxyurea dose in the predicted treatment range, due to potential pitfalls in lab draws, serum storage, sample processing, or hydroxyurea analysis, will start at a default dose of 20.0 ± 2.5 mg/kg/day. For all participants, the hydroxyurea dose will be adjusted as needed based on blood counts to establish the optimal dose. Where necessary, a weekly dosing average will be determined, so that treatment can occur solely with locally available and affordable 500mg hydroxyurea capsules.

SUMMARY:
ADAPT is a prospective cohort study at Jinja Regional Referral Hospital (JRRH) primarily to assess the effect of hydroxyurea on blood transfusion utilization and secondarily to determine the feasibility of PK-guided hydroxyurea dosing.

DETAILED DESCRIPTION:
Hypothesis

* There will be a 50% reduction in the rate of blood transfusions received during the hydroxyurea treatment period compared with the pre-treatment period.
* A PK-guided starting dose will be generated for 80% of participants.
* Participants on PK-guided hydroxyurea treatment will require 25% fewer blood transfusions during their first year of hydroxyurea than those on dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with documented HbSS disease
* Age: ≥ 12 months and ≤ 10 years of age, at the time of enrollment
* Parent or guardian willing and able to provide informed consent
* Able to comply with all study related treatments, evaluations, and follow-up

Exclusion Criteria:

* Current hydroxyurea treatment (or within the past 6 months)
* Regular blood transfusions (6 or more within the past 12 months)
* Transfusion within the last 30 days (temporary exclusion)
* Known malignancy or other known chronic illnesses including but not limited to active tuberculosis, renal disease
* Current participation in other therapeutic clinical trials, or within 6 months of prior disease-modifying treatments

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the rates of blood transfusions overall and by specific indications in children with sickle cell anaemia (SCA), prior to and during hydroxyurea treatment | One year (Enrollment - Month 15)
  The incidence rate ratio of transfusions overall and by specific indication during the screening phase as compared to the treatment phase

SECONDARY OUTCOMES:
To determine clinical and laboratory factors associated with reduction in blood transfusions for children with SCA on hydroxyurea treatment | One year (Enrollment - Month 15)
  The relative risk of transfusion due to the most common clinical diagnoses and laboratory factors for children with SCA on hydroxyurea treatment.

OTHER OUTCOMES:
To assess the feasibility and safety of a pharmacokinetic (PK)-based hydroxyurea dose within the predicted treatment range for Uganda | One year (Enrollment - Month 15)
  The percentage of successful PK-dosing assessments, defined as assessments completed in entirety resulting in the generation of a PK-guided starting dose.
  The incidence rate ratio of clinical and laboratory adverse events among those started on the PK-guided hydroxyurea dose during the screening phase compared with the treatment phase.
To quantify rates of SCA-related complications (including stroke, sepsis, and pain) in participants receiving PK-guided hydroxyurea dosing and within the overall cohort on hydroxyurea treatment | One year (Enrollment - Month 15)
  The number of participants with sickle cell-related complications (including stroke, sepsis and pain) in participants receiving PK-guided hydroxyurea dosing compared to the rate of events in the default dosing group.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Study Director — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Jinja Regional Referral Hospital (JRRH), Department of Paediatrics, Sickle Cell Clinic, Jinja, Uganda

REFERENCES:
- [Derived] Power-Hays A, Namazzi R, Dong M, Kazinga C, Kato C, Aliwuya S, McElhinney K, Conroy AL, Lane A, John C, Vinks AA, Latham T, Opoka RO, Ware RE. The feasibility of pharmacokinetic-based dosing of hydroxyurea for children with sickle cell anaemia in Uganda: Baseline results of the alternative dosing and prevention of transfusions trial. Br J Clin Pharmacol. 2025 Jun;91(6):1865-1872. doi: 10.1111/bcp.70071. PMID 40441700
- [Derived] Power-Hays A, Namazzi R, Dong M, Kazinga C, Kato C, Aliwuya S, McElhinney K, Conroy AL, Lane A, John C, Vinks AA, Latham T, Opoka RO, Ware RE. The feasibility of pharmacokinetic-based dosing of hydroxyurea for children with sickle cell anaemia in Uganda: Baseline results of the alternative dosing and prevention of transfusions trial. Br J Clin Pharmacol. 2025 Apr 13;91(6):1865-72. doi: 10.1002/bcp.70071. Online ahead of print. PMID 40222814